CLINICAL TRIAL: NCT03963934
Title: Feasibility of a Program on a Nurse-led Telephone 6-month-follow-up for Uncontrolled Hypertensive Women: a Patient-tailored Intervention
Brief Title: Feasibility of a Program on a Nurse-led Telephone 6-month-follow-up for Uncontrolled Hypertensive Women
Acronym: PreDynamiques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A01921-56
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Arterial Hypertension; Medication Nonadherence
Keywords: Nurse-led management; Home blood pressure; Nurse-led telephone follow-up
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, open, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with uncontrolled hypertension (Experimental): Women with uncontrolled hypertension and unsatisfactory medication adherence
  Interventions: Other: Program on a nurse-led telephone 6-month-follow-up for uncontrolled hypertensive women: a patient-tailored intervention

INTERVENTIONS:
Other: Program on a nurse-led telephone 6-month-follow-up for uncontrolled hypertensive women: a patient-tailored intervention — Implementation of personalized support: The accompaniment includes 7 telephone interviews for 6 months (understanding the antihypertensive treatment, identifying the brakes and the levers when taking medication, organizing the treatment taking, making the home blood pressure)

SUMMARY:
This study evaluate the feasibility of a 6-month personalized support program for hypertensive and non-observant women, led by nurses by telephone follow-up.

DETAILED DESCRIPTION:
The program includes 2 themes:

1. "Realizing my blood pressure self-measurement" according to the recommendations
2. "Optimizing my compliance": understand the antihypertensive treatment, identify the brakes and the levers when taking medication, organize the treatment taking

Visits :

1. Inclusion visit :

   * Collection of consent by the nurse
   * Verification of inclusion and non-inclusion criteria : measurement of compliance with a scale for each antihypertensive treatment and BP measurement
   * Data collection and goal setting
   * Urine collection for dosing anti-hypertension drugs
   * Delivery of the schedule of telephone visits that were determined with the patient
2. Implementation of personalized support with the following steps :

   * Data collection : evaluate knowledge and its potential as a patient, identify his needs
   * Determination of objectives : define the objectives of the program in each theme with the patient according to the collection of data Implementation of personalized support
   * 7 telephone interviews of 20 to 30 minutes use of specific teaching tools and materials by thematic assessment of achievements, validation of objectives

   Evaluation of the accompaniment:

   - assessment at the final visit
3. Final visit at 6-month : Same as the inclusion visit with assessment of the support and questionnaire to assess the patient satisfaction level.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 to 79 years old,
* Hypertensive and treated with antihypertensive drug(s)
* Unsatisfactory compliance for at least one of her antihypertensive treatment with a score below 80% at the medication adherence scale
* Uncontrolled Blood Pressure (BP) : systolic BP equals to ou greater than140 and / or diastolic BP equals to ou greater than 90 mmHg at inclusion visit
* Inform consent signed
* Affiliation to a French social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Patient with a history of cardio or cerebrovascular disease in the last 6 months (Stroke or Transient Ischemic Attack, myocardial infarction, heart failure)
* Patient with kidney failure requiring dialysis
* Patient with cognitive pathology: dementia, ... etc.
* Patient with type I diabetes
* Unreachable patient by phone or foreseeable inability or unwillingness to comply with study follow-up
* Patient who does not understand and does not speak French

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of women who completed all telephone follow-ups and came to the final visit at 6 months. | 6 months
  The goal of recruitment in 6 months will be 20 women and the goal of the program finalization will be of at least 80% of patients (16 patients).

CONTACTS AND LOCATIONS:
Overall Officials: Edith DAUCHY, RN, Principal Investigator — CHRU Nancy

IPD SHARING:
Plan to Share IPD: No